CLINICAL TRIAL: NCT03900091
Title: Paediatric Infections Point-Of-Care: Point-of-care Approach for Rapid and Easy Meningitis Diagnosis
Brief Title: Paediatric Infections Point-Of-Care
Acronym: PI-POC
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Mbarara University of Science and Technology (Other); Science for Life Laboratory (Unknown); Epicentre Mbarara Research Center (Unknown); Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Tobias Alfvén, Associate Professor, Karolinska Institutet
Other Study IDs: 2018/1676-31/1
Record Dates: First submitted 2019-03-19; First posted 2019-04-02 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Meningitis; Pediatric Infectious Diseases
Keywords: Point of care; Diagnostics; Low-income countries; Meningitis; Pediatrics; MxA; FilmArray; Low-cost diagnostics
MeSH Terms: conditions — Meningitis | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid Nasopharyngeal swabs Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Cases with clinical meningitis: Patients aged 0-12 years with suspected CNS infection, at the pediatric clinics at Mbarara Regional Referral Hospital or Holy Innocents Children's Hospital, Mbarara, Uganda.
  Interventions: Diagnostic Test: Multiplex PCR assay for meningitis; Diagnostic Test: Multiplex vertical flow microarrray assay for meningitis; Diagnostic Test: Profiling of blood proteins by multi-analyte Profiling technology; Other: Typing and whole genome sequencing
- Control subjects: Patients aged 0-12 years, visiting the outpatient pediatric clinics at Mbarara Regional Referral Hospital or Holy Innocents Children's Hospital, Mbarara, Uganda, with fever clinically considered non-severe.
  Interventions: Diagnostic Test: Profiling of blood proteins by multi-analyte Profiling technology; Other: Typing and whole genome sequencing

INTERVENTIONS:
Diagnostic Test: Multiplex PCR assay for meningitis — CSF from cases to be analysed with a FilmArray ME Panel
  Other Names: Biomerieux FilmArray ME Panel
  Groups: Cases with clinical meningitis
Diagnostic Test: Multiplex vertical flow microarrray assay for meningitis — CSF from cases will also undergo analysis with a newly developed prototype for point-of-care diagnostic tool for CNS infections identification. The tool is a DNA-based vertical flow microarray technology printed on paper.
  Groups: Cases with clinical meningitis
Diagnostic Test: Profiling of blood proteins by multi-analyte Profiling technology — Blood from cases and controls to be analysed using Luminex technology to identify protein profiles associated with severe and non-severe infection. Myxovirus protein A (MxA) will also be analysed by the Luminex assay, to associate MxA levels with severe/non-severe infection.
  Other Names: Luminex Multi-Analyte Profiling (xMAP)
Other: Typing and whole genome sequencing — Pathogenic strains isolated from nasopharyngeal swabs from cases and controls will undergo whole genome sequencing (WGS) and typing .

SUMMARY:
This study aims to identify the aetiology of childhood meningitis in Southwestern Uganda and develop and evaluate new methods for point-of-care diagnosis of childhood meningitis in a low-income setting. A prospective observational study including 600 children aged 0-12 years will be conducted during 1 year in Mbarara, Uganda. We estimate to recruit about 300 children with suspected meningitis (cases), and 300 with non-severe infection age-matched as controls.

DETAILED DESCRIPTION:
The current gold standard for laboratory diagnostics of suspected childhood meningitis are microbiology culture of CSF and polymerase chain reaction (PCR). However, these methods are expensive, time-consuming, require dedicated facilities and trained professionals, that are often lacking in low-income health systems. Our team has developed a new vertical flow paper printed microarray method for rapid, inexpensive and multiplexed microbiology analysis of cerebrospinal fluid (CSF), with potential for point-of-care use in low-income settings. This study will evaluate the diagnostic accuracy of this newly developed paper printed microarray method.

The bioMérieux FilmArray® ME Panel is an existing multiplexed PCR based system for rapid microbiology analyses of CSF. Even though previous studies have reported good diagnostic accuracy of the FilmArray® system, the studies have mostly been focused on evaluating the system in high-income settings.

This study will do a field evaluation of the diagnostic performance and clinical usability of the FilmArray® ME Panel in a low-income setting in Mbarara, Uganda.

A study by Page et al, conducted 2009-2012 in Mbarara, Uganda, identified the most frequent pathogen causing childhood bacterial meningitis to be Streptococcus pneumoniae. This is also the case on a global level, with the addition of the bacteria Neisseria meningitidis and Haemophilus influenzae type B. However, the Page study did not find a single case of Neisseria meningitidis, which is in contrast to most other reports from low-, middle- and high-income countries. Furthermore, after the finalisation of the Page study, pneumococcal conjugate vaccines were introduced to the Ugandan childhood immunisation program. This study will identify the current aetiology of childhood meningitis and the impact of the pneumococcal conjugate vaccine, in Mbarara, Uganda, and also study the carriage and characteristics of Neisseria meningitis in children in the area.

Myxovirus resistance protein A (MxA) blood levels have been reported to be elevated in children with respiratory tract infections of viral aetiology, as compared to bacterial aetiology. Previous studies have also shown a higher abundance of MxA in viral encephalitis, however this only through histological analyses of post-mortem brain tissue samples.

This study aims to investigate the correlation of blood MxA levels in children with viral, bacterial and malarial meningitis in Mbarara, Uganda by analysing the protein profile and temporal dynamic in blood of children with severe and non-severe infection.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 months to 12 years of age, who
* meet the case or control definition criteria, and where
* informed consent is obtained from the parent or guardian

Exclusion Criteria:

* all 3 inclusion criteria not met
* No, insufficient or inappropriate CSF sample collection

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: CASE DEFINITION:
  Patients aged 0-12 years, with suspected CNS infection understood as, having fever in the past 48 hours (children <9 months may present with any temp)) AND recent onset of any of the following:
  * Non-traumatic reduced consciousness; in pre-verbals <9 months Blantyre coma score <4; Blantyre coma score <5 for older pre-verbals. In verbal children Glasgow Coma Scale <15
  * prostration, hypotonia/hypertonia, unexplained irritability
  * severe headache
  * photophobia
  * neck stiffness or bulging fontanel
  * seizure(s)
  * focal neurological signs
  * age >18 months: positive Kernig or Brudzinski signs
  * Skin petechiae
  * Cheyne Stokes CNS infection can be suspected for other reasons
  CONTROL DEFINITION:
  Patients aged 0-12 years, visiting the outpatient pediatric clinics with fever and not meeting the case inclusion criteria.
  For every case, one age-matched control will be sought until included.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of vertical flow microarray printed on paper for pathogen identification in human cerebrospinal fluid samples | Patient CSF will be analysed with culture, PCR and FilmArray during ongoing patient management in Mbarara, Uganda. Analyses on frozen patient CSF samples with vertical flow paper printed microarray will be done in Stockholm, Sweden within 1 year.
  The newly developed assay will be evaluated with regards to diagnostic accuracy. For this, results will be compared with those from bacterial culture, PCR and FilmArray analyses of the same samples.

SECONDARY OUTCOMES:
Protein profile variance between children with severe and non-severe infection | Frozen patient blood samples will be analyzed using Luminex Multiplex Assays in Stockholm, Sweden, within 1 year after sample collection in Mbarara, Uganda.
  Protein profile (biomarker) concentration (e.g. μg/L) variance in the blood of children with severe infection as compared to those with uncomplicated infection, as well as longitudinal variance in protein profile during the course of severe infection.
Variance in concentration of MxA in blood of patients with viral vs. non-viral meningitis and non-severe infection. | MxA concentration measurements will be conducted on the Luminex platform on frozen patient blood samples in Stockholm, Sweden, within a year from sample collection.
  Difference in MxA concentration (e.g. μg/L) in peripheral blood of patients with viral/non-viral meningitis and non-severe infection will be studied with the Luminex platform, to identify any feasibility of MxA to be used as a blood biomarker to differentiate between aetiologies of meningitis and to differentiate meningitis to non-severe infection. This in order to assist differential diagnostics in the clinical management of childhood fever.
Diagnostic performance of the FilmArray ME Panel for meningitis diagnostics in children in a low-income setting | FilmArray analyses on fresh patient CSF samples will be conducted immediately after or within 1 day of sample collection.
  Diagnostic accuracy of the FilmArray® (compared to current gold standard methods PCR and culture) for aetiological diagnosis of CNS infections in children. Sensitivity, specificity, positive and negative predictive values, positive and negative likelihood ratios will be calculated for the results from FilmArray analyses on patient CSF samples.
Clinical impact of the FilmArray ME Panel on management of childhood meningits in a low-income setting. | FilmArray analyses on fresh patient CSF samples will be conducted immediately after or within 1 day of sample collection.
  Parameteres including time to laboratory confirmed diagnosis, time to treatment initiation, duration of hospital stay (all in hours/days) and patient mortality will be measured for suspected cases of meningitis whose CSF has been analyzed using the FilmArray® ME panel.
Usability of the FilmArray ME Panel for meningitis diagnostics in children in a low-income setting. | Questionnaires will be handed out and collected from participants continuously during the 1 year duration of patient inclusion.
  A questionnaire will used to gather experiences from health care personnel in Mbarara involved in clinical management of children with suspected meningitis and laboratory personnel in Mbarara conducting FilmArray analyses, in order to study clinical perspectives on the contribution of FilmArray assays to the management of meningitis, in this low-income setting.
Mapping of Neisseria meningitidis carriage and prevalence in children in Mbarara, Uganda | Nasopharyngeal swabs will be collected upon inclusion to the study. Sequencing and serotyping will be done in Stockholm, Sweden, within 1 year after sample collection.
  Whole genome sequencing and serotyping of any strains of N. meningitidis isolated from nasopharyngeal swabs from included children in Mbarara (cases and controls) will be done to understand the local prevalence of N. meningitidis in severe/non-severely ill children in the district.
Etiology of childhood meningitis in the Mbarara district, Uganda. | CSF culture, PCR and FilmArray analyses will be conducted during the 1 year duration of the study, in Mbarara, Uganda.
  Current aetiology of childhood meningitis in the Mbarara district, Uganda, will be studied through culture, PCR and FilmArray analyses of CSF samples from children with suspected meningitis.
The impact of pneumococcal conjugate vaccines on aetiology of childhood meningits in the Mbarara district. | CSF culture, PCR and FilmArray analyses will be conducted during the 1 year duration of the study, in Mbarara, Uganda.
  Comparison of current (post-vaccination era) to prior (pre-vaccination era) aetiology of childhood meningitis. The pneumococcal vaccine was recently included in the Ugandan childhood immunization program, and just prior to this, the aetiology of childhood meningitis in the Mbarara district was reported by Page et al, finding S. pneumoniae to be the most frequent agent causing bacterial meningitis in the district. Has this changed?

CONTACTS AND LOCATIONS:
Overall Officials: Elias Kumbakumba, MD, Principal Investigator — Mbarara University of Science and Technology; Tobias Alfvén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Uganda (2):
  - Holy Innocents Children's Hospital, Mbarara
  - Mbarara Regional Referral Hospital, Mbarara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rasti R, Kumbakumba E, Nanjebe D, Mlotshwa P, Nassejje M, Mzee J, Businge S, Akankwasa G, Nyehangane D, Gantelius J, Boum Y 2nd, Martensson A, Mwanga-Amumpaire J, Alfven T, Gaudenzi G. Clinical utility of the FilmArray(R) meningitis/encephalitis panel in children with suspected central nervous system infection in a low-resource setting - a prospective study in Southwestern Uganda. BMC Infect Dis. 2025 Mar 22;25(1):396. doi: 10.1186/s12879-025-10732-w. PMID 40121439
- [Derived] Gaudenzi G, Kumbakumba E, Rasti R, Nanjebe D, Reu P, Nyehangane D, Martensson A, Nassejje M, Karlsson J, Mzee J, Nilsson P, Businge S, Loh E, Boum Ii Y, Andersson-Svahn H, Gantelius J, Mwanga-Amumpaire J, Alfven T. Point-of-Care Approaches for Meningitis Diagnosis in a Low-Resource Setting (Southwestern Uganda): Observational Cohort Study Protocol of the "PI-POC" Trial. JMIR Res Protoc. 2020 Nov 4;9(11):e21430. doi: 10.2196/21430. PMID 33146628